CLINICAL TRIAL: NCT07138898
Title: Immunosuppressant Management in Rheumatology Patients Undergoing Elective Total Shoulder Arthroplasty
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-00380
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Rheumatic Disease
Keywords: rheumatoid arthritis; psoriatic arthritis; ankylosing spondylitis; systemic lupus erythematosus; juvenile idiopathic arthritis; spondyloarthritis; polymyalgia rheumatica; giant cell arteritis; vasculitis; granulomatosis with polyangiitis; dermatomyositis; polymyositis; inflammatory bowel disease-associated arthritis
MeSH Terms: conditions — Rheumatic Diseases; Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Arthritis, Juvenile; Spondylarthritis; Polymyalgia Rheumatica; Giant Cell Arteritis; Vasculitis; Granulomatosis with Polyangiitis; Dermatomyositis; Polymyositis | interventions — Methotrexate; Sulfasalazine; Hydroxychloroquine; Leflunomide; Azathioprine; Mycophenolic Acid; Cyclosporine; Tacrolimus; Etanercept; Adalimumab; golimumab; Certolizumab Pegol; Infliximab; Rituximab; belimumab; tocilizumab; Interleukin 1 Receptor Antagonist Protein; canakinumab; Abatacept; secukinumab; ixekizumab; bimekizumab; Ustekinumab; guselkumab; risankizumab; tofacitinib; upadacitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard hold (Active Comparator): Patients will follow the standard perioperative immunosuppressant hold protocol based on guidelines from hip and knee arthroplasty literature. The duration of the hold is determined by medication half-life and infection risk considerations. Postoperatively, medications will be restarted approximately 2 weeks after surgery (+/- 2 days), contingent on wound healing and infection status.
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Hydroxychloroquine; Drug: Leflunomide; Drug: Azathioprine; Drug: Mycophenolate; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Etanercept; Drug: Adalimumab; Drug: Golimumab; Drug: Certolizumab; Drug: Infliximab; Biological: Rituximab; Biological: Belimumab; Biological: Tocilizumab; Biological: Anakinra; Biological: Canakinumab; Biological: Abatacept; Biological: Secukinumab; Biological: Ixekizumab; Biological: Bimekizumab; Biological: Ustekinumab; Biological: Guselkumab; Biological: Risankizumab; Drug: Tofacitinib; Drug: Upadacitinib
- Shorter hold (Experimental): Patients will follow an abbreviated immunosuppressant hold protocol, withhold durations modified based on drug pharmacokinetics to allow a shorter preoperative discontinuation period. Medications will be prescribed as usual by the patient's rheumatologist, only adjusting the interval between last preoperative dose and surgery. The rheumatologist will relay the number of weeks/days between the last dose and surgery date. Postoperatively, medications will be restarted approximately 1 week after surgery (+/- 2 days), provided there are no signs of infection or wound healing complications. Route of Administration
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Hydroxychloroquine; Drug: Leflunomide; Drug: Azathioprine; Drug: Mycophenolate; Drug: Cyclosporine; Drug: Tacrolimus; Drug: Etanercept; Drug: Adalimumab; Drug: Golimumab; Drug: Certolizumab; Drug: Infliximab; Biological: Rituximab; Biological: Belimumab; Biological: Tocilizumab; Biological: Anakinra; Biological: Canakinumab; Biological: Abatacept; Biological: Secukinumab; Biological: Ixekizumab; Biological: Bimekizumab; Biological: Ustekinumab; Biological: Guselkumab; Biological: Risankizumab; Drug: Tofacitinib; Drug: Upadacitinib

INTERVENTIONS:
Drug: Methotrexate — Continue throughout perioperative period
Drug: Sulfasalazine — Continue throughout perioperative period
Drug: Hydroxychloroquine — Continue throughout perioperative period
  Other Names: Plaquenil
Drug: Leflunomide — Continue throughout perioperative period
  Other Names: Arava
Drug: Azathioprine — Control group: Withhold the daily dose 1 week prior to surgery Intervention group: Withhold 2 days prior to surgery
  Other Names: Imuran
Drug: Mycophenolate — Control group: Withhold the daily dose 1 week prior to surgery Intervention group: Withhold 2 days prior to surgery
  Other Names: Cellcept
Drug: Cyclosporine — Control group: Withhold the daily dose 1 week prior to surgery Intervention group: Withhold 2 days prior to surgery
Drug: Tacrolimus — Control group: Withhold the daily dose 1 week prior to surgery Intervention group: Withhold 2 days prior to surgery
Drug: Etanercept — Control group: Schedule surgery 2 weeks after last administered dose Intervention group: Schedule surgery 1 week after last administered dose
  Other Names: Enbrel
Drug: Adalimumab — Control group: Schedule surgery 3 weeks after last administered dose Intervention group: Schedule surgery 1 week after last administered dose
  Other Names: Humira
Drug: Golimumab — Control group: Schedule surgery 5 weeks after last administered 4-week subcutaneous dose or 9 weeks after last administered 8-week intravenous dose.
  Intervention group: Schedule surgery 2 weeks after last administered 4-week subcutaneous dose or 4 weeks after last administered 8-week intravenous dose.
  Other Names: Simponi
Drug: Certolizumab — Control group: Schedule surgery 5 weeks after last administered dose. Intervention group: Schedule surgery 2 weeks after last administered dose.
  Other Names: Cimzia
Drug: Infliximab — Control group: Schedule surgery 9 weeks after last administered intravenous dose.
  Intervention group: Schedule surgery 4 weeks after last administered dose.
  Other Names: Remicaide
Biological: Rituximab — Control: Schedule 7 months after last administered dose. Intervention group: Schedule 3 months after last administered dose.
  Other Names: Rituxan
Biological: Belimumab — Control group: Schedule surgery 2 weeks after last administered subcutaneous weekly dose or 5 weeks after last administered 4-week intravenous dose.
  Intervention group: Schedule surgery 1 week after last administered weekly dose or 2 weeks after last administered 4-week dose.
  Other Names: Benlysta
Biological: Tocilizumab — Control group: Schedule surgery 2 weeks after last administered subcutaneous weekly dose or 5 weeks after last administered 4-week intravenous dose.
  Intervention group: Schedule surgery 1 week after last administered weekly dose or 2 weeks after last administered 4-week dose.
  Other Names: Actemra
Biological: Anakinra — Control group: Schedule surgery 2 days after last administered daily dose. Experimental group: Schedule surgery 1 day after last administered daily dose.
  Other Names: Kineret
Biological: Canakinumab — Control group: Schedule surgery 5 weeks after last administered 4-week dose. Intervention group: Schedule surgery 2 weeks after last administered 4-week dose.
  Other Names: Ilaris
Biological: Abatacept — Control group: Schedule surgery 2 weeks after last administered weekly subcutaneous dose or 5 weeks after last administered monthly intravenous dose.
  Intervention group: Schedule surgery 1 week after last administered weekly subcutaneous dose or 2 weeks after last administered monthly intravenous dose.
  Other Names: Orencia
Biological: Secukinumab — Control group: Schedule surgery 5 weeks after last administered subcutaneous dose.
  Intervention group: Schedule surgery 2 weeks after last administered subcutaneous dose.
  Other Names: Cosentyx
Biological: Ixekizumab — Control group: Schedule surgery 5 weeks after last administered 4-week dose. Intervention group: Schedule surgery 2 weeks after last administered 4-week dose.
  Other Names: Taltz
Biological: Bimekizumab — Control group: Schedule surgery 9 weeks after last administered 8-week dose. Intervention group: Schedule surgery 4 weeks after last administered 8-week dose
  Other Names: Bimzelx
Biological: Ustekinumab — Control group: Schedule surgery 13 weeks after last administered 12-week dose. Intervention group: Schedule surgery 6 weeks after last administered 12-week dose.
  Other Names: Stelara
Biological: Guselkumab — Control group: Schedule surgery 9 weeks after last administered 8-week dose. Intervention group: Schedule surgery 4.5 weeks after last administered 8-week dose.
  Other Names: Tremfya
Biological: Risankizumab — Control group: Schedule surgery 13 weeks after last administered 12-week dose. Intervention group: Schedule surgery 6-7 weeks after last administered 12-week dose.
  Other Names: Skyrizi
Drug: Tofacitinib — Control group: Schedule surgery 4 days after last administered daily dose. Intervention group: Schedule surgery 2 days after last administered daily dose.
  Other Names: Xeljanz
Drug: Upadacitinib — Control group: Withhold 4 days prior to surgery Intervention group: Withhold 2 days prior to surgery
  Other Names: Rinvoq

SUMMARY:
The purpose of this study is to assess the incidence of rheumatologic flares, changes in pain scores (VAS), changes in functional outcomes (PROMIS), wound complications, surgical site infections, and return trips to the operating room for rheumatology patients following shoulder replacements, comparing those who stop their immunosuppressants preoperatively for the same amount of time as suggested in the literature for hip and knee arthroplasty versus those who hold the medications for a shorter period of time preoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older at the time of informed consent;
2. Diagnosis of rheumatic disease: rheumatoid arthritis (RA), psoriatic arthritis (PA) , ankylosing spondylitis (AS), systemic lupus erythematosus (SLE), juvenile idiopathic arthritis (JIA), spondyloarthritis, polymyalgia rheumatica, giant cell arteritis, vasculitis, granulomatosis with polyangiitis, dermatomyositis, polymyositis, and inflammatory bowel disease-associated arthritis;
3. On active immunosuppression for at least 3 months prior to scheduled surgery;
4. Scheduled for elective total shoulder arthroplasty;
5. Able and willing to provide written informed consent prior to any study specific procedures.

Exclusion Criteria:

* Patients with active infections or malignancies;
* Patients undergoing shoulder arthroplasty for fracture or tumor;
* Pregnancy or breastfeeding;
* Unable to provide informed consent;
* Patients with severe SLE with marked activity - as they should be offered enrollment in the observational arm. All such patients should remain on treatment to avoid worsening of disease activity;
* Unable or without capacity to provide written informed consent prior to any study specific procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of wound complications | 90-day post operation
Incidence of superficial surgical site infections | 90-day post operation
Incidence of deep surgical site infections | 90-day post operation
Incidence of return trips to the operating room | 90-day post operation
Incidence of rheumatologic disease flares | 90-day post operation

SECONDARY OUTCOMES:
Length of hospital stay | From admission to discharge (on average 2 days)
Postoperative pain score as assessed by the VAS for Pain | Week 2
  Visual Analogue Scale (VAS) for Pain is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Postoperative pain score as assessed by the VAS for Pain | Week 6
  Visual Analogue Scale (VAS) for Pain is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Postoperative pain score as assessed by the VAS for Pain | Month 3
  Visual Analogue Scale (VAS) for Pain is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Change in Range of motion (ROM) - active forward elevation (AFE) | Week 2, Month 3
  The normal range for AFE is between 170 and 180 degrees. A decrease suggests reduced range of motion.
Change in Range of motion (ROM) - external rotation (ER) | Week 2, Month 3
  Normal ER ROM can range from 70 to 90 degrees. A decrease suggests reduced range of motion.
Change in Range of motion (ROM) - internal rotation (IR) | Week 2, Month 3
  The normal IR ROM is 70 to 90 degrees. A decrease suggests reduced range of motion.
Change in PROMIS - Physical Function (PF) - Short Form 10a | Week 2, Month 3
  The PROMIS PF-10a asks respondents to rate their ability to perform 10 physical activities. The responses are summed to create a raw score, which ranges from 10 (representing the lowest level of physical function) to 50 (representing the highest level of physical function).
Change in PROMIS - Pain Interference - Short Form 6a | Week 2, Month 3
  The questionnaire consists of 6 items assessing pain interference. Participants are asked to rate each item from 1 (not at all) to 5 (very much). The PROMIS Pain Interference - Short Form 6a has a possible raw score range of 6 to 30, where higher scores indicate greater pain interference. This raw score is then converted to a T-score, which has a mean of 50 and a standard deviation of 10 in a reference population.
Change in American Shoulder and Elbow Surgeons (ASES) score | Week 2, Month 3
  The ASES questionnaire is a patient-reported outcome measure used to assess shoulder function and pain. It includes a pain scale (using a visual analog scale) and a functional subscale assessing activities of daily living. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Change in Disabilities of the Arm, Shoulder and Hand (DASH) score | Week 2, Month 3
  The DASH is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb. Scores range from 0 to 100, with 0 indicating no disability and 100 indicating the most severe disability. A higher DASH score reflects greater disability and severity of symptoms.
Proportion of participants who used rescue medications or corticosteroid bursts | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Samuels, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: jonathan.samuels@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to jonathan.samuels@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.